**Title:** A double-blinded, placebo-controlled study to evaluate the tolerability and efficacy of Enstilar<sup>®</sup> (calcipotriene and betamethasone dipropionate) Foam in the treatment of chronic plaque psoriasis in patients with skin of color (Fitzpatrick skin phototypes IV-VI).

PI: Andrew Alexis, M.D., MPH

NCT03506477

August 10, 2017

## **Statistical Analysis Plan**

- Categorical outcomes were compared between treatment groups using a 0.05 level Fisher's exact test.
- Continuous outcomes were compared using Wilcoxon signed-rank tests.